CLINICAL TRIAL: NCT05899153
Title: Quantifying Patient-specific Changes in Neuromuscular Control in Cerebral Palsy: Adaptation and Biofeedback During Gait
Brief Title: Gait Adaptation and Biofeedback for Cerebral Palsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Gillette Children's Specialty Healthcare (Other); Northern Arizona University (Other)
Responsible Party: Principal Investigator, Katherine Steele, Professor, Mechanical Engineering, University of Washington
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00015348; R01NS091056 (NIH)
Record Dates: First submitted 2023-05-24; First posted 2023-06-12 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Cerebral Palsy
Keywords: Gait; Rehabilitation
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Orthopedic Surgery (Experimental): Participants who have been scheduled for lower-extremity, multilevel orthopedic surgery will be assessed before and 9-18 months after surgery to evaluate changes in gait and adaptation rates.
  Interventions: Procedure: Multilevel Orthopedic Surgery
- Audiovisual + Sensorimotor Biofeedback (Experimental): Participants will complete 12 sessions (20 minutes of walking on a treadmill) over a 6-8 week period while receiving both audiovisual and sensorimotor biofeedback. Sensorimotor biofeedback will be provided with an ankle exoskeleton that provides resistance to ankle plantarflexion during the stance phase of gait. The visual feedback will be provided on a screen with a bar showing real-time muscle activity and the audio feedback will be a sound played when they reach the target level of muscle activity from the plantarflexors.
  Interventions: Device: Biomotum Spark: Robotic ankle resistance; Device: Audiovisual Biofeedback

INTERVENTIONS:
Device: Biomotum Spark: Robotic ankle resistance — Robotic ankle exoskeleton that provides resistance to ankle plantarflexion.
  Arms: Audiovisual + Sensorimotor Biofeedback
Device: Audiovisual Biofeedback — Electromyography recordings from the plantarflexor muscles are used to provide audio feedback via a sound that plays when muscle activity is above target and a visual bar that displays real-time muscle activity.
  Arms: Audiovisual + Sensorimotor Biofeedback
Procedure: Multilevel Orthopedic Surgery — Musculoskeletal surgeries to address alignment, contracture, and other lower-extremity impairments. This study does not impact surgical decision making but evaluates changes in gait before and after surgery.
  Arms: Orthopedic Surgery

SUMMARY:
This research aims to evaluate walking function in children with cerebral palsy (CP). The researchers want to understand how children with CP adapt and learn new ways of moving. They have previously found that measuring how a person controls their muscles is important for assessing walking ability and response to interventions. In these studies, they will adjust the treadmill belt speeds and/or provide real-time feedback to evaluate how a child can alter their movement. The feedback will include a wearable exoskeleton that provides resistance to the ankle and audio and visual cues based on sensors that record muscle activity. This research will investigate three goals: first, to measure how children with CP adapt their walking; second, to see if either repeated training or orthopedic surgery can improve adaptation rates; and third, to determine if individual differences in adaptation relate to improvements in walking function after treatment. This research will help develop better treatments to enhance walking capacity and performance for children with CP.

DETAILED DESCRIPTION:
Prior research has shown that children with cerebral palsy (CP) use simplified motor control strategies compared to nondisabled (ND) peers, and that these differences in motor control are associated with walking function. While we can quantify motor control during activities like walking, the processes by which a child with CP adapts and learns new movement patterns are poorly understood.

This research will use two paradigms to evaluate adaptation and motor learning in children with CP: walking on a split-belt treadmill and responding to multimodal biofeedback. Walking on a split-belt treadmill, which has two belts set at different speeds to induce asymmetry during walking, has been commonly used to evaluate adaptation in other clinical populations. Responding to multimodal feedback can also be used to evaluate an individual's capacity to adapt their walking pattern. This research will use a real-time multimodal feedback system that targets plantarflexor activity, a key muscle group that is often impaired in CP. Sensorimotor feedback will be provided using a lightweight, body-worn robotic device that provides adaptive ankle resistance and step-by-step audiovisual feedback will be provided based on muscle activity from the plantarflexors using a visual display and audible tone. This research will quantify adaptation rate (e.g., change in soleus activity or step length symmetry) in response to these perturbations, and observe the impact of repeated practice or orthopedic surgery on walking function (e.g., change in walking speed). The specific aims are to:

Aim-1: Quantify adaptation rates in children with CP. We will quantify adaptation rate in response to three perturbation experiments: split-belt treadmill walking, sensorimotor feedback, and audiovisual feedback. The primary hypotheses are that children with CP will exhibit reduced adaptation rates compared to ND peers, and that adaptation rates will be associated with function (Gross Motor Function Measure, GMFM-66).

Aim-2: Determine whether adaptation rates change in response to repeated multimodal feedback training. We will evaluate children with CP who undergo six weeks of multimodal biofeedback training (20-min, 2x/week) or orthopedic surgery. The primary hypothesis is that multimodal feedback training will produce greater changes in adaptation rates than orthopedic surgery.

Aim-3: Determine whether changes in gait after treatment are associated with adaptation rates. Gait analysis will be performed to determine whether baseline adaptation rates are associated with changes in gait after treatment. The primary hypotheses are that baseline adaptation rates will be associated with changes in muscle, joint, and whole-body performance.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bilateral cerebral palsy that impacts both legs
* Gross Motor Functional Classification System Level II
* No surgery or lower-extremity injuries 12 months prior to enrollment
* No botulinum toxin injections in prior 3 months
* No prior selective dorsal rhizotomy surgery
* No history of seizures or cardiac conditions that would preclude walking on a treadmill for 20 minutes
* No current pain that hinders walking

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-11-28 (Actual); Primary Completion 2028-05-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in Soleus Muscle Activity | Change from baseline to intervention follow-up, assessed up to 18 months
  Average stance-phase magnitude of soleus muscle activity from electromyography recording measured during gait at 1-month follow-up.
Change in Peak Ankle Power | Change from baseline to intervention follow-up, assessed up to 18 months
  Average peak ankle power evaluated during gait.
Change in Self-Selected Walking Speed | Change from baseline after intervention.
  Average overground walking speed.
Change in Dynamic Motor Control During Walking (Walk-DMC) | Change from baseline to intervention follow-up, assessed up to 18 months
  The total variance account for by one muscle synergy calculated from electromyography recordings during gait.
Change in Gait Deviation Index (GDI) | Change from baseline to intervention follow-up, assessed up to 18 months
  Deviation in gait kinematics compared to nondisabled gait.
Change in Gross Motor Function Measure - 66 (GMFM-66) Parts D & E | Change from baseline to intervention follow-up, assessed up to 18 months
  Assessment tool designed and evaluated to measure changes in gross motor function. Parts D & E focus on standing, walking, jumping, and running function.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine M Steele, PhD, Principal Investigator — University of Washington
Locations (1):
- Gillette Children's, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data from gait analysis and outcome measures will be provided on a public data repository.
Supporting Information: Study Protocol
Time Frame: Data will be made available within one year after completion of data collection.